CLINICAL TRIAL: NCT04891809
Title: Isatuximab in Combination With Lenalidomide-Dexamethasone Compared to Lenalidomide-Dexamethasone in Elderly Patients (Aged ≥70 Years) With Newly Diagnosed Myeloma: a Randomized Phase II Study (SGZ-2019-12650)
Brief Title: Isatuximab in Combination With Rd Compared to Rd in Elderly Patients (Aged ≥70 Years) With NDMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: University of Navarra (Other); Medical University of Vienna (Other); Assign Data Management and Biostatistics GmbH (Other); WiSP GmbH (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MM-4
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: Myeloma; Isatuximab; Lenalidomide; Dexamethasone; Elderly; age ≥70
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — isatuximab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned in a 1:1 ratio to one of the two arms. Randomization will be stratified by the simplified frailty scale (Facon et al, Leukemia 2020) result nonfrail or frail.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IRd followed by IR (Experimental): Induction: 8 cycles isatuximab+lenalidomide+dexamethasone; Maintenance: up to 24 cylces isatuximab+lenalidomide
  Interventions: Drug: Isatuximab-Irfc 20 MG/ML [Sarclisa]; Drug: Lenalidomide; Drug: Dexamethasone Oral
- Rd followed by R (Other): Induction: 8 cycles lenalidomide+dexamethasone; Maintenance: up to 24 cylces lenalidomide
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Isatuximab-Irfc 20 MG/ML [Sarclisa] — Induction: 10mg/kg on day 1,8,15,22 in cycle 1, subsequently on day 1, 15; every 28 days (q28 days) Maintenance: 10mg/kg, day1, q28 days until progression or intolerance but for a maximum of 24 cycles from start of maintenance
  Arms: IRd followed by IR
Drug: Lenalidomide — Induction: 25mg*, day 1-21, every 28 days (q28 days); Maintenance: 5-10mg, day 1-21, q28 days (according to individual tolerance) until progression or intolerance but for a maximum of 24 cycles from start of maintenance
  *) for patients with moderate renal impairment (30≤ GFR (MDRD formula) < 50 mL/min) starting dose is 10 mg
Drug: Dexamethasone Oral — Induction:
  Patients aged <75 years: 40mg, once weekly; Patients aged ≥75 years: 20mg, once weekly

SUMMARY:
As optimal tolerance is the key for developing new treatments for the very elderly population, the aim of the study is to compare the efficacy and tolerance of isatuximab in combination with lenalidomide+dexamethasone (Rd) versus Rd only in very elderly patients aged 70 years or older. ln sum, a clear and clinically highly relevant benefit is expected with the isatuximab-based triple combination compared to the standard Rd doublet.

DETAILED DESCRIPTION:
The treatment goals in elderly patients with multiple myeloma (MM) are similar to those in younger patients: rapid and long-lasting symptom control, deep response and durable remissions as well as increased survival are at the forefront, similar to therapy goals in younger patients. Elderly patients frequently present with comorbidities, reduced treatment tolerance and greater frequency of treatment discontinuations. Hence, treatment needs to be adapted to the specific needs of this patient population.

ln the recent decade lenalidomide-based therapies have been established as effective treatment modalities in elderly patients. In elderly patients lenalidomide + dexamethasone (Rd) is one of the most frequently used treatment regimens, which is effective and well tolerated.

MM is a high unmet medical need and as a result, several agents are currently under clinical investigation in MM. Monoclonal antibodies (mAb) are one of the most promising groups of drugs in development in the treatment of MM with several of them demonstrating activity in this disease. lsatuximab is a highly effective monoclonal antibody with an excellent activity and tolerance profile, active as single agent therapy in patients with multiple prior lines of treatment.

Presently several trials with isatuximab-lenalidomide containing treatment regimens are ongoing. The expected benefits of adding isatuximab to Rd over Rd alone in very elderly patients seem to outweigh possible risks by far.

A greater depth of response is anticipated including greater number of MRD (minimal residual disease) negative patients, higher response rates, and longer progression free survival.

Risk conferred with the addition of isatuximab are mainly restricted to a roughly 40% rate of infusion reactions, which usually are seen at the first infusion only. ln addition, there is an increased risk for grade 4 leukopenia, grade 2 and 3 thrombocytopenia, and grade 3 infection and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Able to provide written informed consent in accordance with federal, local, and institutional guidelines
* Patients must have newly diagnosed, symptomatic multiple myeloma with evidence of measurable disease (assessed within 21 days prior to randomization)

  * Serum M protein ≥0.5 g/dL measured using serum protein immunoelectrophoresis and/or
  * Urine M protein ≥200 mg/24 hours measured using urine protein immunoelectrophoresis and/or
  * In subjects without detectable serum or urine M-protein, serum free light chain (SFLC) ≥100 mg/L (involved light chain) and an abnormal FLC ratio
* No prior treatment for multiple myeloma
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
* Patients at cardiac risk (NYHA >ll) or pre-existing coronary heart disease, or any other clinically relevant cardiac complication) should be scheduled for a baseline ECHO and can only be included if the LVEF is >40%
* Adequate organ and bone marrow function within the 21 days prior to randomization defined by:

  * Bilirubin < 2 times the upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN
  * absolute neutrophil count (ANC) ≥ 750/mm3 (growth factor support for max 3 days allowed to achieve this value)
  * Hemoglobin >8.0 g/dL (Use of erythropoietic stimulating factors and red blood cell [RBC] transfusion per institutional guidelines is allowed, however the most recent RBC transfusion may not have been done within 7 days prior to obtaining screening hemoglobin.)
  * Platelet count >50,000/mm3
  * Calculated or measured creatinine clearance (CrCl) of ≥30 mL/min; Calculation should be based on the MDRD formula (age, gender, black/non- black, weight, height)

Exclusion Criteria:

* ECOG status >2
* Patients unlikely to tolerate Rd
* Waldenström macroglobulinemia
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia (> 2.0 x 10^9/L circulating plasma cells by standard differential)
* Myelodysplastic syndrome
* Smoldering Myeloma and MGUS
* Second malignancy within the past 5 years except:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Prostate cancer ≤ Gleason score 6 with stable prostate-specific antigen (PSA over 12 months)
  * Ductal breast carcinoma in situ with full surgical resection (i.e., negative margins)
  * Treated medullary or papillary thyroid cancer
  * Other tumors with low risk of recurrence/metastases and/or early stage R0 surgery
* History of or current amyloidosis
* Glucocorticoid therapy within the 14 days prior to randomization that exceeds an accumulated dose of 160 mg dexamethasone or 1000 mg prednisone
* Extended field radio therapy (more than 3 fields) within the 21 days prior to randomization
* Contraindication to isatuximab, dexamethasone, lenalidomide or any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs
* Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, acute diffuse infiltrative pulmonary disease, pericardial disease, or myocardial infarction within 4 months prior to enrolment
* Active infection within the 14 days prior to randomization requiring systemic antibiotics and/or antiviral therapy
* Uncontrolled hypertension or uncontrolled diabetes despite medication
* Significant neuropathy (Grade 2 with pain or Grade 3 or higher) within the 14 days prior to randomization
* Known cirrhosis
* Known human immunodeficiency virus (HIV) seropositivity or active hepatitis C or hepatitis B infection (subjects with past hepatitis B virus [HBV] infection or resolved HBV infection defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti HBc] antibody test are eligible; subjects positive for hepatitis C virus [HCV] antibody are eligible only if polymerase chain reaction [PCR] is negative for HCV RNA.)
* Participation in another interventional study within the 28 days prior to randomization
* Major surgery (except kyphoplasty) within the 28 days prior to randomization
* Any other clinically significant medical disease or social condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent, be compliant with study procedures, or provide accurate information.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with MRD (minimal residual disease) negativity (defined by NGF [next generation flow] at 10^-5) after end of induction treatment in the two arms. | After 8 months of induction treatment (8 cycles, each cyle is 28 days)
  To demonstrate the benefit of isatuximab in combination with lenalidomide and low-dose dexamethasone followed by isatuximab and lenalidomide maintenance therapy in changing the proportion of patients with MRD negativity as compared to lenalidomide and low-dose dexamethasone followed by lenalidomide maintenance treatment in patients with newly diagnosed multiple myeloma (NDMM).

SECONDARY OUTCOMES:
Percentage of patients with response to study treatment | After 32 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment)
  Effect of treatment on Overall Response Rate (ORR) including patients with Partial Response (PR), Very Good Partial Response (VGPR) and Complete Response (CR) as per International Myeloma Working Group (IMWG) criteria in each arm.
Progression-free Survival | After 44 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment and a minimum of 12 months of follow-up)
  Effectiveness of treatments on Progression-free survival (PFS)
Overall Survival | After 44 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment and a minimum of 12 months of follow-up)
  Effectiveness of treatments on Overall Survival (OS)
Effectiveness of treatments on MRD negativity | After 20 months (8 months of induction treatment and 12 months of maintenance treatemnent)
  To evaluate the proportion of patients with MRD negativity (defined by NGF [next generation flow] at 10^-5) after 12 months (13 cycles) of maintenance treatment.
Effectiveness of treatments on preventing progressive disease | After 44 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment and a minimum of 12 months of follow-up)
  To evaluate the Time to Progression (TTP) in each arm.
Progression-free Survival in different high-risk cytogenetic populations | After 44 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment and a minimum of 12 months of follow-up)
  Effectiveness of treatment on PFS in high risk cytogenetic populations defined as patients carrying a) del(17p), t(4;14), t(14;16) in each arm and b) the same aberrations plus amp1q21.
Duration of response | After 44 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment and a minimum of 12 months of follow-up)
  Length of time between response and progression or death.
Incidence of treatment-emergent adverse events (Safety and tolerability) | After 32 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment)
  Number of participants with treatment-emergent adverse events as assessed by NCI-CTCAE Version 5.0.
Changes in quality of life (QoL) using general questionnaire European Organization for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ) Core 30 (C 30) (EORTC-QLQ-C30) | After 32 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment)
  Changes in quality of life will be analyzed by using the cancer patient-specific questionnaire EORTC-QLQ-C30.
Changes of general health status using questionnaire EQ (EuroQol) 5 dimension (5D) 5 level (5L) (EQ-5D-5L) | After 32 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment)
  Changes in general health status will be analyzed by using the questionnaires EQ-5D-5L. QoL.
Changes in quality of life (QoL) using multiple myeloma specific questionnaire EORTC-QLQ Myeloma (MY) 20 (EORTC-QLQ-MY20) | After 32 months (8 months of induction treatment and a maximum of 24 months of maintenance treatment)
  Changes in quality of life will be analyzed by using the multiple myeloma-specific questionnaire EORTC-QLQ-MY20.
Progression-free survival after second line therapy | After end of study treatment until 12 months of follow up as a minimum (until LPLV)
  Influence of potential second line therapy on Progression-free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, Principal Investigator — Wilhelminen Cancer Research Institute, Clinic Ottakring
Locations (14):
- Austria (9):
  - Bezirkskrankenhaus Kufstein, Innere Medizin, Interne II u. onkologische Tagesklinik, Kufstein
  - LKH Hochsteiermark - Leoben, Abt. f. Innere Medizin, Haemato-Onkologie, Leoben
  - Univ.Klinikum Krems, Klin. Abt. f. Innere Medizin 2, Mitterweng
  - PMU Salzburg: Universitätsklinik für Innere Medizin III, Salzburg
  - Univ.-Klinikum St. Pölten, Innere Medizin 1, Sankt Pölten
  - Krankenhaus d. Barmh. Schwestern Wien, 1. Med. Abteilung, Onkologie und Hämatologie, Vienna
  - Hanusch Krankenhaus der Österreichischen Gesundheitskasse, 3. Med. Abteilung, Vienna
  - Klinik Ottakring, 1.Med.Abt., Zentrum f. Onkologie, Haematologie und Palliativmedizin, Vienna
  - Krankenhaus Zams, Innere Medizin, Internistische Onkologie-Haematologie, Zams
- Greece (3):
  - General Hospital of Athens "Evangelismos", Hematology Clinic, Athens
  - General Hospital of Athens "Alexandra, Plasma Cell Dyscrasias Unit, Athens
  - Anticancer Hospital of Thessaloniki "Theageneio", Hematology, Thessaloniki
- Serbia (2):
  - University Clinical Center of Serbia, Clinic for Hematology, Belgrade
  - University Clinical Center Kragujevac, Clinic for Hematology, Kragujevac

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Facon T, Dimopoulos MA, Meuleman N, Belch A, Mohty M, Chen WM, Kim K, Zamagni E, Rodriguez-Otero P, Renwick W, Rose C, Tempescul A, Boyle E, Manier S, Attal M, Moreau P, Macro M, Leleu X, Lorraine Chretien M, Ludwig H, Guo S, Sturniolo M, Tinel A, Silvia Monzini M, Costa B, Houck V, Hulin C, Yves Mary J. A simplified frailty scale predicts outcomes in transplant-ineligible patients with newly diagnosed multiple myeloma treated in the FIRST (MM-020) trial. Leukemia. 2020 Jan;34(1):224-233. doi: 10.1038/s41375-019-0539-0. Epub 2019 Aug 19. PMID 31427722
- See also: Sponsor — http://www.agmt.at